CLINICAL TRIAL: NCT07085195
Title: A Clinical Study of the Safety and Efficacy of Chemogenetics Therapy in the Treatment of Parkinson's Disease
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Chemogenetics
Record Dates: First submitted 2025-07-15; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Parkinson Disease (PD); Gene Therapy; Safety and Efficacy; Clozapine
MeSH Terms: conditions — Parkinson Disease | interventions — Genetic Therapy; Clozapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- all of 6 patients plan to receive chemogenetic gene therapy (Experimental): This is a single-arm and open-label study design for initial safety assessment. Six participants will be divided into three dose groups in the dose escalation principle. The dose escalation principle is as follows:
  After the first sentinel subject receives 1×10¹² vg virus vector, the research team will evaluate the safety, tolerability, and efficacy of the current drug dose after 4 weeks. If this sentinel does not experience dose-limiting toxicity, another sentinel subject will receive a 2×10¹² vg dose; if this sentinel develops dose-limiting toxicity (DLT), this dose will be defined as an intolerable dose, and the Data Review Committee will determine whether to select a lower dose for exploration or terminate dose escalation based on the existing data. If this sentinel subject doesn't experience dose-limiting toxicity, another subject will receive 4×10¹² vg dose. If this sentinel subject doesn't experience DLT, all of the next three subjects will receive 4×10¹² vg dose.
  Interventions: Genetic: gene therapy; Drug: clozapine

INTERVENTIONS:
Genetic: gene therapy — Six participants are planned to be divided into three dose groups in the dose escalation principle. The dose escalation principle is as follows: After the first sentinel subject receives 1×10¹² vg virus vectors, the research team will evaluate the safety, tolerability, and efficacy of the current drug dose after 4 weeks. If this sentinel does not experience dose-limiting toxicity, another sentinel subject will receive a 2×10¹² vg dose; if this sentinel develops dose-limiting toxicity (DLT), this dose will be defined as an intolerable dose, and the Data Review Committee will determine whether to select a lower dose for exploration or terminate dose escalation based on the existing data. If this sentinel subject doesn't experience dose-limiting toxicity, another participant will receive a 4×10¹² vg dose as a new sentinel subject. If this sentinel subject doesn't experience DLT, all of the next three subjects will receive a 4×10¹² vg dose.
Drug: clozapine — Clozapine ramp-up will be performed four weeks after neurosurgery, when the participants have recovered, and the participants will be treated orally with clozapine. Clozapine is 25mg per tablet, and the oral dose is 1/32, 1/16, and 1/8 tablet twice a day, in the morning and at noon, respectively, with each dose repeated for 3 days for a total of 9 days. If no DLT develops during this time, the participants will continue to take 1/8 pill orally twice a day as a maintenance dose, and they will be monitored for 12 months.

SUMMARY:
The investigators propose a gene therapy strategy using chemical genetic inhibition to intervene in the abnormal activity of the subthalamic nucleus in Parkinson's disease. The investigators design and construct a highly efficient therapeutic injection STP-001 (first drug), through the efficient adeno-associated virus capsid (AAV), neuronal promoter (hSyn), and chemical genetic effector element (hM4Di), and accurately inject the drug into the bilateral subthalamic nucleus, the core pathological nucleus of Parkinson's disease, through stereotactic technology. Combined with a very low dose of clozapine (the second drug), the abnormal activity of the subthalamic nucleus is precisely intervened to improve the core motor symptoms of Parkinson's disease.

DETAILED DESCRIPTION:
This is a single-arm and open-label study design for initial safety assessment. 6 cases of patients with iPD will be recruited from the neurology department of Ruijin Hospital, Affiliated Shanghai Jiao Tong University, School of Medicine. After the informed consent is signed, six participants will be divided into three dose groups in the dose escalation principle to receive the STP-001 injection. The virus dose escalation principle is as follows:

After the first sentinel subject receives 1×10¹² vg virus vectors, the research team will evaluate the safety, tolerability, and efficacy of the current drug dose after 4 weeks. If this sentinel does not experience dose-limiting toxicity, another sentinel subject will receive a 2×10¹² vg dose; if this sentinel develops dose-limiting toxicity (DLT), this dose will be defined as an intolerable dose, and the Data Review Committee will determine whether to select a lower dose for exploration or terminate dose escalation based on the existing data. If this sentinel subject doesn't experience dose-limiting toxicity, another subject will receive a 4×10¹² vg dose. If this sentinel subject doesn't experience DLT, all of the next three subjects will receive a 4×10¹² vg dose. 4 weeks After receiving the STP-001 injection, when the participants have recovered, clozapine ramp-up will be performed, and the participants will be treated orally with clozapine. Clozapine is 25 mg per tablet, and the oral dose is 1/32, 1/16, and 1/8 tablet twice a day, in the morning and at noon, respectively, with each dose repeated for 3 days for a total of 9 days. If no DLT develops during this time, the participants will continue to take 1/8 pill orally twice a day as a maintenance dose, and they will be monitored for 12 months.

ELIGIBILITY:
Inclusion criteria

Participants who meet all the following criteria can be included in this clinical study:

1. Clinically diagnosed with idiopathic Parkinson's Disease [in accordance with the Diagnostic Criteria for Parkinson's Disease in China published in 2016, or in accordance with the Diagnostic Criteria for Primary PD of the International Parkinson's and Movement Disorders Society (MDS) in 2015];
2. Subjects aged 40-65 years old (including the boundary value), regardless of gender;
3. Medical history of disease ≥5 years;
4. Hoehn-Yahr staging scale for "off" period is 2.5-4;
5. Regular use of dopaminergic drugs before the screening period, including taking levodopa for at least 4 weeks;
6. MDS-UPDRS III score >35 in the "off" period, and the improvement rate of acute levodopa stress test ≥30%;
7. AAV neutralizing antibody titer ≤1:2000;
8. The subject agrees to postpone other neurosurgery during the main study phase (including deep brain stimulation, except for sudden life-threatening conditions requiring neurosurgery during the trial);
9. No acute adverse reactions to the scheduled therapeutic dose of clozapine (1-month observation period);
10. The subject agrees not to participate in other therapeutic intervention studies during the trial;
11. The subject agrees not to be vaccinated during the study phase;
12. Use reliable contraceptive methods from the screening period to at least 8 weeks after drug infusion;
13. The subject has good compliance and can follow up regularly. During the follow-up period, the PD patient diary can be accurately completed. Family members, guardians, or caregivers can help the subject fill in the patient diary;
14. The subject fully understands the nature, purpose, methods, and possible adverse reactions of this clinical trial, voluntarily participates as a subject, and signs the informed consent form; if the subject is unable to read, the legal agent or impartial witness can read the informed consent form and other written materials and witness the informed consent.

Exclusion criteria

If any of the following criteria are met, the patient shall be excluded from this study:

1. Atypical or secondary Parkinson's syndrome (such as Parkinson's plus syndrome, hereditary Parkinson's syndrome, drug-induced Parkinson's syndrome);
2. Contraindications to surgery or previous deep brain stimulation surgery, pallidotomy, extrapyramidal surgery, other brain surgeries, or other neurosurgery that the researcher determines will affect their participation in this trial;
3. Previous cranial imaging suggests abnormal brain structure, cerebrovascular malformations, intracranial tumors, intracranial hemorrhage risk, brain trauma, and other abnormalities;
4. Mini-Mental State Examination (MMSE) score <24 points;
5. Montreal Cognitive Assessment (MoCA) score <26 points;
6. Mini-Mental State Questionnaire (PHQ-9) ≥16;
7. Abnormal liver and kidney function: Aspartate aminotransferase (AST) or Alanine aminotransferase (ALT) > 1.5 times the upper limit of normal value, serum creatinine (Cr) >1.5 times the upper limit of normal value;
8. Abnormal coagulation function or using anticoagulants;
9. Infectious disease screening: Hepatitis B surface antigen (HBsAg) or hepatitis B virus DNA (HBV-DNA) positive, hepatitis C virus RNA (HCV-RNA) positive, human immunodeficiency virus (HIV) positive, or syphilis serum positive;
10. Undergoing antiviral treatment for hepatitis B and hepatitis C;
11. Suffering from unstable or severe other systemic diseases: including active tuberculosis, cardiovascular system, respiratory system, Diseases of the digestive system, urinary system, mental and nervous system (such as epilepsy), blood system, immune system, etc., or abnormal laboratory test values, the investigator determines that the patient is not suitable for participating in this trial;
12. Suffering from malignant tumors or having a history of malignant tumors;
13. Having had severe allergic reactions, allergic to contrast agents, or being unable to accept surgical anesthesia;
14. Participating in other clinical trials or having participated in other clinical trials within 3 months before the screening period;
15. Having received gene therapy before being enrolled into this trial;
16. Having received stem cell therapy within 6 months before the screening period;
17. Having used other investigational drugs within 4 weeks before screening or within 5 half-lives of the investigational drug (whichever is longer), or drugs that the investigator determines affect this trial;
18. Having received live vaccines within 2 months before the screening period or having a history of vaccination within 30 days before the screening period;
19. Have a history of alcohol dependence or drug addiction and cannot stop drinking as advised by the doctor during the trial;
20. Female subjects who are pregnant or breastfeeding;
21. Severe motor complications after anti-PD drug treatment and no suitable alternative treatment options;
22. Subjects who are assessed by the researchers as unsuitable for inclusion.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
1. The incidence of adverse events and serious adverse events within 12 months after bilateral subthalamic nucleus injection of STP-001, which is the adeno-associated virus vector carrying the target gene. | Electrocardiogram and laboratory tests will be conducted at baseline and then prior to, during, and after the neurosurgery operation and 4, 12, 24, 36, and 48 weeks after administration of the intervention.
  Adverse events and serious adverse events will be assessed by electrocardiogram and laboratory tests for safety and tolerability assessment, including routine blood tests, routine urine tests, and blood biochemistry.
2. The changes in the titer levels of the binding and capsid-neutralizing antibodies against adeno-associated virus in serum within 12 months after bilateral subthalamic nucleus injection of STP-001. | The titer levels of binding and capsid-neutralizing antibodies will be conducted at baseline, at the time after the neurosurgery operation, and at 12, 24, 36, and 48 weeks after administration of the intervention.
  The changes in the titer levels of the binding and capsid-neutralizing antibodies against adeno-associated virus in serum will be assessed for safety and tolerability assessment.

SECONDARY OUTCOMES:
The differences of anti-PD drug usage before and after treatment | The anti-PD drug usage will be conducted at baseline, at the time after the neurosurgery operation, and at 12, 24, 36, and 48 weeks.
  Compare the changes in anti-PD drug use, including daily oral levodopa or a levodopa-equivalent dose, from baseline to post-treatment in 6 participants.
The differences of the MDS-Unified Parkinson's Disease Rating Scale before and after treatment | 12, 24, 36, and 48 weeks
  Compare the changes in the MDS-Unified Parkinson's Disease Rating Scale from baseline to post- treatment in all of the 6 participants.
The differences of the Patient Global Impression improvement scale before and after treatment | 12, 24, 36, and 48 weeks
  Compare the changes in the Patient Global Impression improvement scale from baseline to post-treatment in all of the 6 participants.
The differences of the Clinical Global Impression scale-improvement before and after treatment | 12, 24, 36, and 48 weeks
  Compare the changes in the Clinical Global Impression scale-improvement from baseline to post-treatment in all of the 6 participants
The differences of the Gait and Falls questionnaires before and after treatment | 12, 24, 36, and 48 weeks
  Compare the changes in the Gait and Falls questionnaires from baseline to post-treatment in all of the 6 participants.
The differences of the Non-Motor Symptoms Questionnaire before and after treatment | 12, 24, 36, and 48 weeks
  Compare the changes in the Non-Motor Symptoms Questionnaire from baseline to post-treatment in all of the 6 participants.
The differences of the Scales for Outcomes in Parkinson's Disease Autonomic before and after treatment | 12, 24, 36, and 48 weeks
  Compare the changes in the Scales for Outcomes in Parkinson's Disease Autonomic from baseline to post-treatment in all of the 6 participants.
The differences of the REM Sleep Behavior Disorder Screening Questionnaire before and after treatment | 12, 24, 36, and 48 weeks
  Compare the changes in the REM Sleep Behavior Disorder Screening Questionnaire from baseline to post-treatment in all of the 6 participants.
The differences of the Sniffin' Sticks 16-item Test and Pittsburgh Sleep Quality Index before and after treatment | 12, 24, 36, and 48 weeks
  Compare the changes in the Sniffin' Sticks 16-item Test and Pittsburgh Sleep Quality Index from baseline to post-treatment in all of the 6 participants.
The differences of the Montreal Cognitive Assessment and Mini-Mental State Examination before and after treatment | 12, 24, 36, and 48 weeks
  Compare the changes in the Montreal Cognitive Assessment and Mini-Mental State Examination from baseline to post-treatment in all of the 6 participants.
The differences of the Mini-Mental State Examination before and after treatment | 12, 24, 36, and 48 weeks
  Compare the changes in the Mini-Mental State Examination from baseline to post-treatment in all of the 6 participants.
The differences of the Hamilton Depression Scale before and after treatment | 12, 24, 36, and 48 weeks
  Compare the changes in the Hamilton Depression Scale from baseline to post-treatment in all of the 6 participants.
The differences of the Hamilton Anxiety Scale before and after treatment | 12, 24, 36, and 48 weeks
  Compare the changes in the Hamilton Anxiety Scale from baseline to post-treatment in all of the 6 participants.
The differences of the Parkinson's Disease Sleep Scale-2 before and after treatment | 12, 24, 36, and 48 weeks
  Compare the changes in the Parkinson's Disease Sleep Scale-2 from baseline to post-treatment in all of the 6 participants.
The differences of the Parkinson's Disease Questionnaire before and after treatment | 12, 24, 36, and 48 weeks
  Compare the changes in the Parkinson's Disease Questionnaire from baseline to post-treatment in all of the 6 participants.
The differences of the Tinetti Performance Oriented Mobility Assessment before and after treatment | 12, 24, 36, and 48 weeks
  Compare the changes in the Tinetti Performance Oriented Mobility Assessment from baseline to post-treatment in all of the 6 participants.
The differences of the Berg balance scale before and after treatment | 12, 24, 36, and 48 weeks
  Compare the changes in the Berg balance scale from baseline to post-treatment in 6 participants.
The differences of the Webster Rating Scale before and after treatment | 12, 24, 36, and 48 weeks
  Compare the changes in the Webster Rating Scale from baseline to post-treatment in 6 participants.
The changes of the MRI before and after treatment | 12, 24, 36, and 48 weeks
  Compare the changes in the MRI examination, including BOLD-MRI, DTI, QSM, and NM-MRI, from baseline to post-treatment in 6 participants.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of neurology, Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: No